CLINICAL TRIAL: NCT05299112
Title: An Exploratory Study of Increased Preterm Arginine INTake on Biological Pathways Affecting Immune Function in Infants Requiring Early Parenteral Nutrition
Brief Title: An Exploratory Study of Increased Preterm Arginine INTake (PAINT18)
Acronym: PAINT18
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool Women's NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LWH1213
Record Dates: First submitted 2022-02-15; First posted 2022-03-28 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Preterm; Nutritional Deficiency; Immune System and Related Disorders
Keywords: Preterm; Arginine; Immune function; Nutrition
MeSH Terms: conditions — Premature Birth; Malnutrition | interventions — Arginine

STUDY DESIGN:
Intervention Model Description: There will be parallel assignment of supplemented parenteral nutrition (PN) and standard parenteral nutrition dependent upon stock availability of intervention PN.
Masking Description: This is not blinded or randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard parenteral nutrition (No Intervention): These infants will form the control group and will receive standard parenteral nutrition. They will be sub-stratified into infants <27 weeks and infants >27 weeks gestation.
- Arginine supplementation (Experimental): These infants will form the intervention group and will receive parenteral nutrition with additional arginine (18% of amino acid) for up to 14 days of life. They will be sub-stratified into infants <27 weeks and infants >27 weeks gestation.
  Interventions: Dietary Supplement: Arginine

INTERVENTIONS:
Dietary Supplement: Arginine — The intervention parenteral nutrition contains additional arginine (18% arginine content) as compared to standard parenteral nutrition (6.3% arginine content).
  Arms: Arginine supplementation

SUMMARY:
PAINT18 is a nutrition study focusing on the effect of arginine supplementation on immune function in preterm infants.

The investigators will explore the effect of current intravenous feeding (parenteral nutrition (PN) formulations on blood arginine levels and the genes that are involved in body nutrition and fighting infection in premature babies. The investigators will also investigate the effect of supplementing arginine on these genes. The investigators will undertake a single centre exploratory physiological study in 24 very premature infants receiving PN. 16 of these infants will be supplemented with arginine. The investigators will record nutritional intake and routine biochemical testing data (which includes amino acid levels) collected over the first 30 days of life. The investigators will take blood for analysis at prespecified intervals for RNA sequencing, ammonia and IGF-1 levels. RNA sequencing findings will allow the investigators to describe the effect of arginine on gene activity in preterm infants

The investigators hypothesise that arginine supplementation will result in changes in gene expression that are consistent with changes in T-cell function and associated inflammatory pathways.

DETAILED DESCRIPTION:
Title The effect of increased Preterm Arginine INTake on biological pathways affecting immune function in infants requiring early parenteral nutrition (PAINT-18 )

Population Preterm infants <29 weeks gestation and/or <1200g

Number of infants 24 infants (completing the study) will be recruited over approximately 12 months

Number of sites One. Infants will be born at Liverpool Women's Hospital (LWH) or transferred to LWH within 48 hours of birth.

Study duration Informed consent will take place antenatally, where possible, or within 72 hours of birth. The first study related blood sample will be taken on day 3 of life with the last sample taken on day 30 of life. Other study assessments reflect those routinely performed in preterm infants receiving parenteral nutrition (PN).

Study intervention All infants will receive standard clinical treatment. 8 infants will receive PN with Vaminolact as the amino acid base, with 6.3% arginine content, and 16 infants will receive PN with additional arginine in the PN bag at a concentration of 18%. These 16 infants will be sub-stratified into two groups based on gestational age (23-26 weeks and 27-29 weeks).

Primary objective To examine the changes in gene expression present in arginine supplemented infants <29 weeks' gestation and/or <1200g between day 3 and day 10 of life. This will be done via illumina RNA sequencing and statistical pathway analysis. The changes in gene expression will be compared with those seen between day 3 and day 10 in unsupplemented infants. The genes of interest are those involved in immune function and inflammatory pathways. Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.

Secondary objectives

1. To examine the changes in gene expression present in arginine supplemented infants <29 weeks' gestation and/or <1200g between days 3, 10 and day 30 of life. This will be done via illumina RNA sequencing and statistical pathway analysis. The changes in gene expression will be compared with those seen between days 3, 10 and day 30 in unsupplemented infants. The genes of interest are those involved in immune function and inflammatory pathways. Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.
2. Statistical pathway analysis will be used to identify genes and their relationship with key biological pathways i) known to be involved in the pathogenesis of necrotising enterocolitis ii) involved in arginine metabolism iii) that are related to the insulin-IGF-I axis
3. To compare the changes in metabolomic profiles of control and intervention infants during the first 30 days of life.
4. To compare growth (weight and head circumference) and body composition data including total body water (intracellular and extracellular distribution) and fat free mass during study period

ELIGIBILITY:
Inclusion Criteria:

* Infants born <29 weeks' gestation
* and/or with birthweight <1200g
* Admitted to the Neonatal Unit at Liverpool Women's Hospital within 48 hours of birth.

Exclusion Criteria:

* Infants who are unlikely to survive the first week after birth.
* Infants known (or suspected to have) a diagnosis of inborn error of metabolism or serious liver dysfunction
* Parents who are unable to give informed consent

Ages: 22 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Gene expression via Illumina RNA sequencing | Day 3 and 10 of life
  RNA will be extracted from whole blood and sent for Illumina RNA sequencing. These sequences are then mapped to reference gene sets for gene expression analysis. The pattern of alteration in gene expression between days 3 and 10 in arginine deficient preterm infants after correction of their deficiency by supplementation with arginine will be analysed. The changes in gene expression will be compared with those seen in unsupplemented infants. The genes of interest are those involved in T-cell function and associated inflammatory pathways. Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.

SECONDARY OUTCOMES:
Gene expression via Illumina RNA sequencing | Days 3, 10 and 30 of life
  RNA will be extracted from whole blood and sent for Illumina RNA sequencing. These sequences are then mapped to reference gene sets for gene expression analysis. The pattern of alteration in gene expression between days 3, 10 and 30 in arginine deficient preterm infants after correction of their deficiency by supplementation with arginine will be analysed. The changes in gene expression will be compared with those seen in unsupplemented infants. The genes of interest are those involved in T-cell function and associated inflammatory pathways. Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.
  Secondary analysis will include Day 30 measurements.
Gene expression via Illumina RNA sequencing | Day 3, 10 and 30 of life
  RNA will be extracted from whole blood and sent for Illumina RNA sequencing. These sequences are then mapped to reference gene sets for gene expression analysis. The pattern of alteration in gene expression between days 3, 10 and 30 in arginine deficient preterm infants after correction of their deficiency by supplementation with arginine will be analysed. The changes in gene expression will be compared with those seen in unsupplemented infants. The genes of interest are those known to be associated with necrotising enterocolitis (NEC). Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.
Gene expression via Illumina RNA sequencing | Day 3, 10 and 30 of life
  RNA will be extracted from whole blood and sent for Illumina RNA sequencing. These sequences are then mapped to reference gene sets for gene expression analysis. The pattern of alteration in gene expression between days 3, 10 and 30 in arginine deficient preterm infants after correction of their deficiency by supplementation with arginine will be analysed. The changes in gene expression will be compared with those seen in unsupplemented infants. The genes of interest are those known to be involved with arginine metabolism. Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.
Blood ammonia levels | Day 3, 10 and 30 of life
  Blood ammonia levels will be measured at day 3, 10 and 30 of life and levels in supplemented intervention infants will be compared to unsupplemented control infants.
Plasma arginine levels | Day 3, 10 and 30 of life
  Plasma arginine levels will be measured at day 3, 10 and 30 of life and levels in supplemented intervention infants will be compared to unsupplemented control infants.
Plasma proline levels | Day 3, 10 and 30 of life
  Proline is a urea cycle intermediate involved in arginine metabolism. Plasma proline levels will be measured at day 3, 10 and 30 of life. Metabolomics profiling and analysis will be used to compare supplemented intervention infants with unsupplemented control infants.
Body composition measuring total body fluid measured in litres | Day 3, 10 and 30 of life
  Body composition measurements will be taken regularly via bioelectrical impedance measuring total body fluid (intracellular and extra cellular distribution) during the study period. Results from control and intervention infants will be compared.
Body composition measuring fat free mass in grams | Day 3, 10 and 30 of life
  Body composition measurements will be taken regularly via bioelectrical impedance measuring fat free mass during the study period. Results from control and intervention infants will be compared.
Growth measuring body weight in grams | Day 3, 10 and 30
  Infants will be weighed regularly during the study period. Measurements from control and intervention infants will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Women's Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available